CLINICAL TRIAL: NCT02439502
Title: Single Center, Prospective, Open Label Post Marketing Study of EndoChoice's Fuse® Endoscopic System Performance In Routine Practice
Brief Title: EndoChoice's Fuse® Endoscopic System Performance In Routine Practice
Acronym: Fuse®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EndoChoice Innovation Center, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CD 1978
Record Dates: First submitted 2015-04-16; First posted 2015-05-08 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Miscellaneous Gastroenterology and Urology Devices Associated With Adverse Incidents, Not Elsewhere Classified

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): Upper and Lower digestive tract diagnostic. The Fuse® system is intended for diagnostic visualization of the digestive tract. The system also provides access for therapeutic interventions using standard endoscopy tools. Fuse Colonoscopies are indicated for use within the lower digestive tract (including the anus, rectum, sigmoid colon, colon and ileocecal valve) for adult subjects and for the upper digestive tract (including the esophagus, stomach, and duodenum).
  Interventions: Device: Fuse® system

INTERVENTIONS:
Device: Fuse® system — Fuse® system will be used to perform gastro and endoscopic diagnostic procedures for upper and lower GI tract.

SUMMARY:
The intent of this study is to evaluate the performance and usability of Fuse in routine practice. The participants are indicated for upper (gastroscopy) and lower (colonoscopy) gastrointestinal endoscopy procedures. The study is open label, prospective and Post Marketing study.

DETAILED DESCRIPTION:
The intent of this study is to evaluate the performance and usability of Fuse in routine practice EndoChoice's Fuse system - Fuse is an FDA, CE and AMAR approved Endoscopic system (Gastroscope and Colonoscope).

Fuse® system The Fuse system is intended for diagnostic visualization of the digestive tract. The system also provides access for therapeutic interventions using standard endoscopy tools. The Fuse system consists of camera heads, endoscopes, video system, light source and other ancillary equipment.

Fuse Colonoscopes in conjunction with the FuseBox™ processor are indicated for use within the lower digestive tract (including the anus, rectum, sigmoid colon, colon and ileocecal valve) for adult subjects.

Fuse Gastroscopes in conjunction with the FuseBox™ processor are indicated for use within the upper digestive tract (including the esophagus, stomach, and duodenum).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18 at least
* The subject has been scheduled for routine screening upper or lower endoscopy, diagnostic work up, or endoscopic surveillance.
* Signed informed consent

Exclusion Criteria:

* Subjects who are currently enrolled in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of findings (abnormal GI findings, such as polyps and tec.) per diagnostic procedure, using Fuse® system | 1 outpatient hospitalization day for subject

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dickstein, MD, Principal Investigator — Carmel Medical Center, Haifa, Israel.